CLINICAL TRIAL: NCT01488760
Title: Deep Abdominal Wall Muscle Dysfunction During Calm Respiration in Chronic Low Back Pain Patients
Brief Title: Abdominal Wall Evaluation in Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FRACINI
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Abnormally Decreased Muscle Contraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Nineteen women with low back pain
- Twenty pain-free women

SUMMARY:
The purpose of this study was to evaluate feed-forward contraction of the transversus abdominis and thickness of the transversus abdominis, obliquus internus, and obliquus externus during calm and standardized respiration in low back pain patients and pain-free subjects.

DETAILED DESCRIPTION:
Low back pain patients have alterations in abdominal wall function, especially in the feed-forward activation of transversus muscle during limbs movements. However, there are no reports on the abdominal function in low back pain patients during physiological respiratory movement.

ELIGIBILITY:
Inclusion Criteria:

* For the low back pain group: women with history of non-specific chronic low back pain for more than three months
* For the pain-free group: pain-free women

Exclusion Criteria:

* For both groups were: pregnancy, neurological condition, obesity (body mass index: BMI >30), or previous spine or abdominal surgery.
* For the low back pain group: rheumatology diseases other than low back pain.
* For the pain-free group: any rheumatology disease.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clarice Tanaka, PhD, Principal Investigator — Full Professor - Department of Physical Therapy, Communication Science & Disorders, Occupational Therapy, Faculty of Medicine - USP; Patricia R Patarro, Study Chair — Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, Brazil; Renato A Sernik, Study Chair — Institute of Radiology, School of Medicine: University of São Paulo, Brazil; Débora M Meira, Study Chair — Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, Brazil; América C Fracini, Study Chair — Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, Brazil; Cássio M Siqueira, Study Chair — Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, Brazil
Locations (1):
- Physical Therapy, Speech and Occupational Therapy Department, School of Medicine: University of São Paulo, Brazil, São Paulo, São Paulo, Brazil